CLINICAL TRIAL: NCT02311296
Title: Effect of Bacterial Colonization and Extracellular HSP-70 Expression in Sub-Glottic Secretions on Ventilator Free Days in Patients Receiving Mechanical Ventilation for Respiratory Failure or Airway Protection
Brief Title: Reduced Ventilator-Free Days and Bacterial Colonization of Sub-Glottic Secretions
Status: Withdrawn | Type: Observational
Why Stopped: Study registered to wrong sponsor.
Sponsor: University of Tennessee, Chattanooga (Other)
Responsible Party: Sponsor
Other Study IDs: HI-LO Study
Record Dates: First submitted 2014-05-13; First posted 2014-12-08 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ventilator associated pneumonia (VAP) is common problem among ICU patients and major source of infection among patients receiving mechanical ventilation. Patients on mechanical ventilation accumulate secretion leading to aspiration of infected secretions. Using new generation endotracheal tube (Hi-Lo tube) can reduce the incidence of VAP.

DETAILED DESCRIPTION:
All patients secrete fluids into the upper airway from the base of our tongue and other related structures. These "subglottic" secretions are normally cleared by swallowing, but when a person requires mechanical ventilation that process is blocked by the breathing tube and the subglottic secretions tend to accumulate. The removal of these subglottic secretions is very important because bacteria that normally inhabit the back of our throats can enter and ultimately colonize collected pools of subglottic secretions. This process is called "micro-aspiration" and has been shown to be strong risk factor for the development of Ventilator associated pneumonia (VAP). Previously, doctors and nurses would attempt to limit these secretions by passing small suction tubes through the breathing tube, but this was found to be ineffective and increased the risk for bleeding and lung injury.

A new development in the management of patients requiring mechanical ventilation is the Hi-Lo endotracheal tube. This device has "suction ports" on either side of the tube that allow for the removal of accumulated subglottic secretions.The standard of care is to use this Hi-Lo ET tube and to remove subglottic secretions every 4-6 hours. The Hi-Lo tube is designed to minimize any suction related trauma. Moreover, recent studies of this ET tube have shown that regular suctioning reduces the incidence of VAP. When these "colonized" secretions were treated with antibiotics, it reduced the number of VAP and shortened the time on the breathing machine. The observation that treatment of bacterial colonization of subglottic secretions reduced the time on the breathing machine is potentially very important clinically. In this study, we propose that the development of bacterial colonization directly contributes to respiratory failure and leads to longer times on the ventilator. The primary aim of the study could lead to reduce the time that patients need mechanical ventilation.

Recent studies have identified a group of "protective proteins" called the heat shock proteins (HSP) that appear to protect patients from developing pneumonia. The protective effect of these proteins is even more pronounced in patients that require mechanical ventilation. Under stressed conditions, HSPs are secreted or released into the subglottic secretions and the level of secretion is sufficient appears to prevent bacteria from "colonizing" the upper respiratory tract.

In addition to looking at rates of bacterial colonization of these secretions, a portion of these secretions to measure the amount of HSP and whether reduced secretion leads to prolonged time on the ventilator.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. Patients requiring mechanical ventilation for altered mental status, drug overdose or any condition that airway protection from aspiration is clinically warranted
3. Patients requiring mechanical ventilation following Cardiothoracic bypass or valve replacement surgery
4. Patients requiring mechanical ventilation for stroke, intra-cranial bleed, sub-dural hematoma, meningitis or closed head injury
5. Patients requiring mechanical ventilation for following of abdominal surgery in which there were no discernable infiltrates on chest X-ray
6. Patients requiring mechanical ventilation for primary lung disease (COPD, emphysema etc.) if no discernable infiltrates on chest X-ray.

Exclusion Criteria:

* 1) Patients receiving mechanical ventilation for greater than 6 hrs at the time of enrollment.

  2) Patients requiring mechanical ventilation for ARDS, pneumonia or traumatic lung injury.

  3) Patients receiving more than one dose of any antibiotic.

  4) Patients undergoing surgical resection for lung cancer or any other surgery directly involving lung parenchyma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
To determine time course and incidence of bacterial colonization of subglottic secretions | first 72 hours of receiving mechanical ventilation

SECONDARY OUTCOMES:
Patients with bacterial colony counts greater than Log(10)4 after 72 hours | after 72 hours of ventilation have reduction of ventilator free days at Day 14

OTHER OUTCOMES:
Secretion of HSP-70 into subglottic secretions | through Day 14
  To determine if secretion of HSP-70 into subglottic secretions of patients with mechanical ventilation reduces the number of patients developing bacterial colonization exceeding Log(10)4 colony forming units/ml

CONTACTS AND LOCATIONS:
Overall Officials: John Gunter, MD, Principal Investigator — University of Tennessee, Chattanooga
Locations (1):
- Erlanger Hospital, Chattanooga, Tennessee, United States